CLINICAL TRIAL: NCT02171442
Title: Metabolism and Pharmacokinetics of [14C]-BIBR 953 ZW After Administration of Single Doses of 5 mg [14C]-BIBR 953 ZW Intravenously or 200 mg [14C]-BIBR 1048 Oral Solution in a Group Comparison Design in 12 Healthy Male Volunteers.
Brief Title: Metabolism and Pharmacokinetics of [14C]-BIBR 953 ZW After Administration of Single Doses of [14C]-BIBR 953 ZW Intravenously or [14C]-BIBR 1048 Oral Solution in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.6
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

ARMS (2):
- BIBR 953 ZW Intravenously (Experimental)
  Interventions: Drug: BIBR 953 ZW Intravenously
- BIBR 1048 Oral Solution (Active Comparator)
  Interventions: Drug: BIBR 1048 Oral Solution

INTERVENTIONS:
Drug: BIBR 953 ZW Intravenously — 5 mg, 2.8 MBq (76 µCi)
  Arms: BIBR 953 ZW Intravenously
Drug: BIBR 1048 Oral Solution — 200 mg free base, 2.8 MBq (76 µCi)
  Arms: BIBR 1048 Oral Solution

SUMMARY:
The aim of this study were to investigate the metabolism and pharmacokinetics of BIBR 1048 MS and BIBR 953 ZW in man.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent from each subject in accordance with the regulatory and legal requirements of the UK
* Age between 30 and 55 years of age
* Body Mass Index (BMI) of between 18.5 and 29.9 kg/m²

Exclusion Criteria:

* Any of the findings from the medical examination (including BP, pulse rate and ECG) deviated from normal or were of clinical relevance
* History of current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of relevant orthostatic hypotension, fainting spells and blackouts, or volunteers with diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the principal investigator
* History of any bleeding disorder including prolonged or habitual bleeding
* History of other hematologic disease
* History of cerebral bleeding (e.g. after a car accident)
* History of craniocerebral trauma
* Intake of drugs with a long half life (≥ 24h) within 1 month prior to administration
* Any drugs which may have had an influence on the results of the trial within 10 days prior to administration or during the trial
* Any volunteers who had participated in another trial with an investigational drug within 3 months ( 4 months if the drug was a new chemical entity) prior to administration or during the trial
* Exposition to radiation in the previous 12 months (i.e. serial x-rays, CT scan or barium meal)
* Smoker
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 12 weeks prior to administration or during the trial
* Any excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of familial bleeding disorder
* Platelets > 150 x 10-9 /l
* Unable to defecate at least once a day every two days

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2002-04; Primary Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Total radioactivity in plasma and whole blood | 168 hours
Total radioactivity in urine and faeces (excretion balance) over 168 h or until < 1% excreted in urine/faeces samples in a 24 h period | over 168 hours or 24 hour period
Concentrations of BIBR 953 ZW in plasma over 168 h, estimation of the extent of gastrointestinal absorption | 168 hours
Concentrations of BIBR 953 ZW in urine | 168 hours
[14C] metabolic pattern and identification of metabolites in urine and if feasible, in plasma and faeces in comparison with various animal species | -12, 0 hours, 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168 post dose

SECONDARY OUTCOMES:
Ratio of radioactivity in blood cells and plasma (CE/CP) | 0.5, 1, 2 ,4 ,8, 24 hours after oral study drug administration, 31min, 1, 2, 4, 8, 24h after start of infusion
Measurement of in vitro plasma protein binding of [14C]-BIBR 953 ZW | Screening, day-1, day 1-day 8
Cmax - Peak (maximum) plasma concentration of BIBR 953 ZW | Screening, day-1, day 1-day 8
tmax - time to reach the peak plasma concentration of BIBR 953 ZW | Screening, day-1, day 1-day 8
t1/2 - Terminal half-life derived from non-compartmental analysis of BIBR 953 ZW | Screening, day-1, day 1-day 8
AUC0-t - area under the plasma concentration vs. time curve from time zero to the time point for the last sample on the pharmacokinetic profile in which total radioactivity or active drug were reliably quantified) BIBR 953 ZW | Screening, day-1, day 1-day 8
AUC0-infinity - Area under the plasma concentration vs. time curve from time zero to infinity - BIBR 953 ZW | Screening, day-1, day 1-day 8
MRT0-inf - the average amount of time a particle remains in a compartment or system, derived when the drug concentration profile is extrapolated to infinity) - BIBR 953 ZW | Screening, day-1, day 1-day 8
MRT0-t - the average amount of time a particle remains in a compartment or system - BIBR 953 ZW | Screening, day-1, day 1-day 8
CL renal - the apparent volume of the central compartment cleared of drug via renal excretion into the urine, per unit time - BIBR 953 ZW | Screening, day-1, day 1-day 8
CLtot - the apparent volume of the central compartment cleared of drug per unit tim after intravenous dosing - BIBR 953 ZW | Screening, day-1, day 1-day 8
CLtot/F - the apparent volume of the central compartment cleared of drug per unit time after extravascular dosing - BIBR 953 ZW | Screening, day-1, day 1-day 8
Vss - apparent volume of distribution at steady state following intravenous administration - BIBR 953 ZW | Screening, day-1, day 1-day 8
Vz/f - Volume of distribution during terminal phase after oral administration - BIBR 953 ZW | Screening, day-1, day 1-day 8
Cmax - Peak (maximum) plasma concentration for total radioactivity | up to day 8
tmax - time to reach the peak plasma concentration for total radioactivity | up to day 8
Occurence of Adverse events | Screening, upt to 10 days after study drug administration
Change from Baseline in physical examination | Screening, 8 to 10 days after study drug administration
Changes from Baseline in vital signs | Screening, 8 to 10 days after study drug administration
Change from Baseline in systolic and diastolic blood pressure | Screening, Day-1, day1, day2, day 8-10 after study drug administration
Change from Baseline in Pulse rate | Screening, Day-1, day1, day2, day 8-10 after study drug administration
Change from Baseline in 12-lead electrocardiogram (ECG) | Screening, Day-1, day1, day2, day 8-10 after study drug administration
Change from Baseline in clinical laboratory tests (hematology, clinical chemistry and urinanalysis) | Screening, day-1, day1, day2, day3, day 8-10 after study drug administration
Changes from baseline in activated partial thromboplastin time - aPTT | Screening, 1, 2, 24, 48 and 168 hours post dose administration
Changes from baseline in coagulation parameter INR - international normalized ratio prothrombin time | Screening, 1, 2, 24, 48 and 168 hours post dose administration